CLINICAL TRIAL: NCT00915473
Title: Greater Occipital Nerve Block for Migraine Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: David W. Dodick M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-008203; UL1TR000135 (NIH)
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Bupivacaine; Saline Solution; Methylprednisolone; Methylprednisolone Hemisuccinate; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Injection (Experimental): Subjects randomized to this arm will receive 2.5 mL 0.5% bupivicaine plus 0.5 mL 20 mg methylprednisolone injected over the ipsilateral (unilateral headache) or bilateral (bilateral headache) occipital nerve.
  Interventions: Drug: bupivicaine; Drug: methylprednisolone
- Placebo Injection (Placebo Comparator): Subjects randomized to this arm will receive 2.75 mL normal saline plus 0.25 mL 1% lidocaine injected over the ipsilateral (unilateral headache) or bilateral (bilateral headache) occipital nerve.
  Interventions: Drug: normal saline; Drug: lidocaine

INTERVENTIONS:
Drug: bupivicaine — 2.5 mL 0.5% bupivicaine
  Other Names: Marcain; Marcaine; Sensorcaine; Vivacaine
  Arms: Active Injection
Drug: normal saline — 2.75 mL normal saline
  Arms: Placebo Injection
Drug: methylprednisolone — 0.5 mL 20 mg methylprednisolone
  Other Names: Medrol; Solu-Medrol
  Arms: Active Injection
Drug: lidocaine — 0.25 mL 1% lidocaine
  Other Names: xylocaine
  Arms: Placebo Injection

SUMMARY:
Migraine is a common neurological condition that can be disabling, particularly if chronic. Greater occipital nerve (GON) block has been utilized for decades for the treatment of migraine in the absence of a single randomized, placebo-controlled trial documenting its effectiveness.

Hypothesis: Greater occipital nerve block reduces the frequency of days with moderate or severe headache in patients with episodic or chronic migraine.

DETAILED DESCRIPTION:
Migraine is a common disease with lifetime prevalence in women and men of 33% and 12% respectively. Chronic migraine affects 2% of the US population and is highly disabling. There are no FDA approved medications for the treatment of chronic migraine.

Although some patients benefit from a daily prophylactic medication, others continue to suffer from severe, frequent, debilitating headaches. Limited efficacy, poor compliance, side effects and drug-drug interactions may explain why more than 80% of migraineurs in the population are not prescribed daily prophylactic medications.

Occipital nerve injections with corticosteroids and/or local anesthetics have been employed for the acute and prophylactic treatment of migraine, cervicogenic headache and cluster headache for decades. A long-acting anesthetic and corticosteroid are often combined, although anesthetic agents have also been used alone. However, there are no randomized controlled trials evaluating the preventive efficacy of occipital nerve block in subjects with migraine.

Patients were equally randomized to receive either 2.5 ml 0.5% bupivacaine plus 0.5 ml 20 mg methylprednisolone over the ipsilateral (unilateral headache) or bilateral (bilateral headache) occipital nerve or 2.75 ml normal saline plus 0.25 ml 1% lidocaine without epinephrine (placebo). The GON injection site was at the medial third of the distance between the occipital protuberance and the mastoid process. Patients were evaluated after the 4-week baseline diary completion phase to undergo the injection, and for 4 weeks after the injection. Therefore, there were 3 patient visits in this study: screening, injection and 4-week follow-up. In an effort to ensure adequate blinding, 0.25 ml of short-acting 1% lidocaine without epinephrine was used as the placebo arm. In order to ensure adequate blinding of the investigator, each syringe and needle hub was covered with opaque tape so as to ensure blinding of the investigator providing the injection. A total of four investigators provided injections. The blinded investigator who evaluated the study subject 4 weeks after injection may or may not be the same as the investigator who provided the injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet diagnostic criteria for episodic migraine or chronic migraine according to the International Headache Classification II (ICHD-II)
* Migraine sufferers who experience at least 1 attack per week
* Able to read and understand the requirements of the study, abide by any restrictions, and return for the required examinations
* Able and willing to sign an informed consent statement
* Subjects must be in generally good health as confirmed by medical history, medication review, baseline physical examination, vital signs and clinical laboratory evaluations.

Exclusion Criteria:

* Subjects with continuous headache (no headache free periods)
* Subjects using maintenance opioid medication
* Subjects who have started a medication with prophylactic migraine efficacy within the past 2 months
* Known hypersensitivity or allergic reaction to any of study ingredients (lidocaine, bupivicaine, any local anesthetics, and corticosteroids) or betadine.
* Use of any investigational medication within 90 days of the initial screening visit and/or concurrent enrolment in an investigational study
* Injection site infection or systemic infection at the injection visit (afebrile at time of injection)
* Presence of cranial bone defect
* Subjects with chronic cluster headache, new daily persistent headache, hemicrania continua, or chronic tension type headache
* Subjects with a history of an unstable medical condition (e.g. cardiovascular, hepatic, renal, endocrine) that may impair their reliable participation in the study or necessitate the use of medications not permitted in this study
* Subjects with a history (within the past 6 months) of a major psychiatric disorder that in the opinion of the investigator may preclude the subject from completed the requirements of the study
* Female subjects who are pregnant or nursing
* Subjects with a history of drug or alcohol abuse within the past 2 years
* Subjects with a history of poor compliance with past drug therapies, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Dodick, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Dilli E, Halker R, Vargas B, Hentz J, Radam T, Rogers R, Dodick D. Occipital nerve block for the short-term preventive treatment of migraine: A randomized, double-blinded, placebo-controlled study. Cephalalgia. 2015 Oct;35(11):959-68. doi: 10.1177/0333102414561872. Epub 2014 Dec 12. PMID 25505035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by referral from multiple neurologists in the division of Headache at Mayo Clinic in Arizona from June 2009 to October 2012.
Period: Screening
Arm/Group | Active Injection | Placebo Injection
Started | 35 | 35
Completed | 34 | 35
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Injection
Arm/Group | Active Injection | Placebo Injection
Started | 34 | 35
Completed | 34 | 35
Not Completed | 0 | 0
Period: 4-week Follow Up
Arm/Group | Active Injection | Placebo Injection
Started | 34 | 35
Completed | 33 | 30
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Injection | Placebo Injection | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 43 (15) | 43 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least 50% Reduction in the Frequency of Days With Moderate or Severe Migraine in the 4 Week Post Injection Compared to the 4 Week Pre-injection Baseline Period
Description: The baseline frequency will be the number of calendar days with moderate or severe migraine during the 4 week period prior to injection, and the follow-up frequency will be the number of calendar days with migraine during the 4 week period following injection.
Time Frame: 4 weeks pre-injection baseline, 4 weeks post-injection
Population: Because of missing data, 33 subjects in the active arm and 30 subjects in the placebo arm were analyzed.
Measure: Number; unit: participants
Arm/Group | Active Injection | Placebo Injection
Number analyzed (Participants) | 33 | 30
participants | 10 | 9
Statistical Analysis 1: Comparison: Active Injection vs Placebo Injection; Test type: Superiority or Other; p = 0.98, Chi-squared

2. Secondary Outcome: Mean Frequency of Days With a Migraine
Time Frame: 4 weeks post-injection
Population: Because of missing data, 33 subjects in the active arm and 30 subjects in the placebo arm were analyzed.
Measure: Mean (Standard Deviation); unit: days per 4 weeks
Arm/Group | Active Injection | Placebo Injection
Number analyzed (Participants) | 33 | 30
days per 4 weeks
  Severe | 3.4 (3.4) | 2.9 (2.7)
  At Least Moderate | 7.0 (4.2) | 7.8 (5.8)
  At Least Mild | 9.3 (4.8) | 10.4 (6.8)
Statistical Analysis 1: Comparison: Active Injection vs Placebo Injection; Severe Migraine Frequency; Test type: Superiority or Other; p = 0.52, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Injection vs Placebo Injection; At least Moderate Migraine Frequency; Test type: Superiority or Other; p = 0.52, t-test, 2 sided
Statistical Analysis 3: Comparison: Active Injection vs Placebo Injection; At Least Mild Migraine Frequency; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

3. Secondary Outcome: Mean Number of Hours With Moderate or Severe Migraine
Time Frame: 4 weeks post-injection
Population: Because of missing data, 33 subjects in the active arm and 30 subjects in the placebo arm were analyzed.
Measure: Mean (Standard Deviation); unit: hours per 4 weeks
Arm/Group | Active Injection | Placebo Injection
Number analyzed (Participants) | 33 | 30
hours per 4 weeks | 60 (72) | 58 (60)
Statistical Analysis 1: Comparison: Active Injection vs Placebo Injection; Test type: Superiority or Other; p = 0.90, t-test, 2 sided

4. Secondary Outcome: Mean Number of Days With Acute Medication Use
Description: Acute medication use meant "the consumption of a drug to abort or terminate a headache."
Time Frame: 4 weeks post-injection
Population: Because of missing data, 33 subjects in the active arm and 30 subjects in the placebo arm were analyzed.
Measure: Mean (Standard Deviation); unit: days per 4 weeks
Arm/Group | Active Injection | Placebo Injection
Number analyzed (Participants) | 33 | 30
days per 4 weeks | 6.7 (4.2) | 7.7 (6.3)
Statistical Analysis 1: Comparison: Active Injection vs Placebo Injection; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events for 4 weeks.
Groups:
- Active Injection: Subjects randomized to this arm will receive 2.5 mL 0.5% bupivicaine plus 0.5 mL 20 mg methylprednisolone injected over the greater occipital nerve.
- Placebo Injection: Subjects randomized to this arm will receive 2.75 mL normal saline plus 0.25 mL 1% lidocaine injected over the greater occipital nerve.
Arm/Group | Active Injection | Placebo Injection
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/35
Other Adverse Events (participants affected / at risk) | 7/34 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Injection (N=34) | Placebo Injection (N=35)
Benign Intracranial Hypertension (pseudotumor cerebri) (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Injection (N=34) | Placebo Injection (N=35)
Injection Site Pain (Onset < or = 1 day) (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Abdominal Distension (Bloating, onset <1 day) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fat Redistribution (onset 22 days) (General disorders) | 1 (1) | 0 (0)
Injection Site Paraesthesia (onset 14 days) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuralgia (Occipital nerve tenderness, onset 61 days) (Nervous system disorders) | 1 (1) | 0 (0)
Weight Increased (onset < 1 day) (General disorders) | 1 (1) | 0 (0)
Fatigue (onset 1 day) (General disorders) | 0 (0) | 1 (1)
Hypoesthesia (numbness) (onset <1 day) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lymphadenopathy (swelling axilla, onset 1 day) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myalgia (Upper extremity muscle soreness, onset 1 day) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (onset 32 days) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (Unspecified, onset 2 days) (General disorders) | 0 (0) | 1 (1)
Pain of Skin (Scalp tenderness, onset < 1 day) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No